CLINICAL TRIAL: NCT01178749
Title: Exploration of Symptom Experience and Related Factors for Patients With Chronic Hepatitis C Infection Receiving 24-week Interferon-α With Ribavirin Treatments: Development of a Prediction Model
Brief Title: Exploration of Chronic Hepatitis C Infection Receiving 24-week Interferon-α With Ribavirin Treatments
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Shiow-Ching Shun / Assistant Professor, National Taiwan University
Other Study IDs: 200708003R
Record Dates: First submitted 2010-04-11; First posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C; Interferon; Symptom Distress; Quality of Life
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic Hepatitis C Infection: patients Receiving 24-week Interferon-α with Ribavirin Treatments

SUMMARY:
The aims of this three-year study are to explore symptom experience and its related factors for the patients with chronic hepatitis C Infection receiving interferon-α with ribavirin for 24 weeks and further to predict the relative risk of failure or occurence of severe side effects which interrupt the treatment.

DETAILED DESCRIPTION:
The antiviral treatment, interferon-α with ribavirin, has been used in treating chronic hepatitis C patients to prevent the development of liver cirrhosis and hepatocellular carcinoma. However, the duration of this treatment needs at least 6 months and severe side effects such as anemia, fatigue, depression with suicidal thoughts can occur at any time throughout the treatment. There has been no study related to the issue of the risk to the population of developing these severe side effects and failing the treatment. Therefore, the aims of this three-year study are to explore symptom experience and its related factors for the patients with chronic hepatitis C Infection receiving interferon-α with ribavirin for 24 weeks and further to develop a prediction model for individuals to predict the relative risk of failure or occurence of severe side effects which interrupt the treatment. Patients will be recruited from outpatients in two hospitals in Northern and Middle Taiwan. A longitudinal study is designed with a one-year follow-up at pre-treatment, and at the 1, 2, 4, 6, 8, 12,16,20, 24 weeks during treatment, and at the 4, 12, 24 weeks of post-treatment. The basic information including the laboratory data, the Symptom Distress Scale, the Fatigue Symptom Inventory, the Hospital Anxiety and Depression Scale, MOS, and the Short-Form 12 Health-Related Quality of Life questionnaires will be used to assess patients' demographic characteristics, symptom experience, fatigue, depression, anxiety, sleep disturbance, and quality of life during the treatment. Three hundred patients will be interviewed within three years. The data will be analyzed using descriptive, independent t-test, Pearson's correlation, Analysis of Variances, generalized estimating equations, logistic regression, and classification tree. We expect this study to explore the characteristics of the population with high risks of treatment failure to severe side effects during treatment in Taiwan. In addition, the results can provide the information for clinicians and researchers to tailor interventions to individual needs.

ELIGIBILITY:
Inclusion Criteria:

* patients with Chronic Hepatitis C Infection Receiving 24-week Interferon-α with Ribavirin Treatments
* Those Who willing to participate in the research
* Aged above 18

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Hepatitis C inpatients
Sampling Method: Non-Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
symptom distress Scale | 6 months
Fatigue symptom inventory | 6 months
The SF-12 health survey | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shiow-Ching Last, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan